CLINICAL TRIAL: NCT02397304
Title: Influence of Pre- or Post-exercise Food Intake on Muscle Metabolism in Obesity
Brief Title: Nutrition, Exercise and Muscle Metabolism in Obesity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Birmingham (Other)
Collaborators: Allen Foundation Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: RG_15-036
Record Dates: First submitted 2015-03-12; First posted 2015-03-24 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Obesity
Keywords: Intra-muscular triglyceride use
MeSH Terms: conditions — Obesity | interventions — Exercise

ARMS (2):
- Pre-exercise food (Experimental): Pre-exercise food provision
  Interventions: Other: Exercise
- Post-exercise food (Experimental): Post-exercise food provision
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — Participants will complete two morning exercise sessions. One will be performed in the overnight fasted-state (i.e. no food or drink, except water, from 10pm the evening before) and the other will be performed in the fed-state having received a breakfast by the research team before exercise.

SUMMARY:
Obesity is a major public health issue and its association with insulin resistance greatly increases risks for cardiovascular disease and type 2 diabetes. Exercise training is recommended for obese populations, but longitudinal studies indicate aerobic exercise training in obese individuals in the absence of weight loss has minimal impact on insulin resistance. High turnover of fat stored within muscle cells (i.e., intramyocellular triglyceride) during exercise and elevated muscle fitness (i.e., muscle oxidative capacity) are key features of the enhanced insulin sensitivity observed in endurance-trained individuals. It could be that longitudinal studies of exercise training in obese individuals failed to sufficiently stimulate intramyocellular triglyceride turnover during exercise and muscle oxidative adaptation as a result of failure to consider the impact of recent nutrition within their study designs. Performing exercise in the fed vs. fasted state can blunt these exercise responses in non-obese individuals. The researchers will investigate the hypothesis that an acute bout of aerobic exercise performed in the overnight-fasted versus fed-state can stimulate greater intramyocellular triglyceride utilization during exercise and enhanced expression of genes related to muscle oxidative adaptation in obese individuals. The expected outcomes will help to determine if exercising in the fasted state could be used to optimise metabolic adaptation to training in obese individuals. The future impact of this research could be the recommendation of a simple nutritional strategy considering meal timing to enhance the effects of aerobic exercise training in obese individuals, with potential long-term benefits for reducing insulin resistance and cardio-metabolic disease risk.

DETAILED DESCRIPTION:
Two thirds of the adult US population is overweight or obese and the prevention and treatment of obesity is a key priority due to the strain on societal health, well-being and economic prosperity. Obesity is associated with insulin resistance characterized by a reduced ability of insulin to stimulate glucose uptake into skeletal muscle and by hyperglycaemia. Obesity and insulin resistance are major risk factors for cardiovascular disease and type 2 diabetes. Weight loss through caloric restriction and increasing physical activity levels are the mainstay of non-surgical/pharmacological treatment for obesity. Weight loss can reduce insulin resistance although sustainable weight loss is difficult to achieve. Physical activity can help with weight maintenance but perhaps surprisingly, carefully controlled longitudinal studies in obese patients indicate aerobic exercise training in the absence of weight loss has no or at best modest impact on peripheral insulin resistance.

One mechanism by which regular aerobic exercise training ensures high peripheral insulin sensitivity in endurance trained individuals is via stimulation of intramyocellular triglyceride turnover and muscle fat oxidation, which maintains low muscle levels of fatty acid metabolites known to interfere with insulin-stimulated muscle glucose uptake (e.g., fatty acyl CoA, diacyglycerols, ceramides). Indirect evidence suggests intramyocellular triglyceride can be utilized as fuel during aerobic exercise in obese individuals, at least in the overnight-fasted state. However, the influence of overnight-fasted vs. fed-state exercise on intramyocellular triglyceride utilization and muscle oxidative adaptation has not been studied in obesity. This is important to study as fed-state exercise, as compared to overnight-fasted exercise, blunts exercise-associated increases in intramyocellular triglyceride utilization, oxidative gene expression, long-term adaptation of muscle oxidative capacity and resistance to high fat diet induced impairments in oral glucose tolerance in lean individuals.

Thus, the presence or timing of recent nutrition with respect to exercise could be a critical factor explaining the inability of aerobic exercise training per se to improve peripheral insulin sensitivity in longitudinal studies in obese populations. Exercising in the overnight-fasted state could optimize metabolic adaptation to training in obese individuals with long-term benefits for reduced insulin resistance and cardio-metabolic disease risk.

ELIGIBILITY:
* Anthropometry/Body Size:

  i. Overweight (White European populations, BMI 25-29.9 kg/m2 or Asian populations, BMI 23-27.4 kg/m2) and have a high waist circumference (European, Sub-Saharan Africans and Eastern Mediterranean and middle east [Arab] men ≥ 94 cm [37 inches], women ≥ 80 cm [31.5 inches]; South Asian, Chinese, Japanese, and ethnic south and central Americans men ≥ 90 cm [35 inches], women ≥ 80 cm [31.5 inches]) or ii. Class I obesity (White European populations, BMI 30-34.9 kg/m2 or Asian populations, BMI 27.5-35 kg/m2).
* Weight stable i.e. (±2 kg) for >3 months before enrolment
* Sedentary i.e. no regular engagement in physical activity
* Diagnosis and general health: Good general health defined as no known cardiovascular or metabolic disease
* Compliance: understands and is willing, able and likely to comply with all study procedures and restrictions
* Consent: demonstrates understanding of the study and willingness to participate as evidenced by voluntary written informed consent.

Exclusion Criteria:

* Answering "YES" to any question on the Screening Form
* Hypertension (≥140/90 mmHg)
* Any ECG Abnormalities
* Current participation in another clinical study
* Current or recent smoker (last 30 days)
* Past history of substance abuse, engagement in uncommon eating practices (e.g., sustained periods of fasting) and taking prescription or non-prescription medication (e.g., beta-blockers, insulin or thyroxine) or supplements that may influence normal metabolic responses.
* Participants who have previously (within 5 years of the present study) had 4 or more muscle biopsies obtained from the thigh quadriceps region will be ineligible

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Estimated)
Dates: Start 2015-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Intramuscular triglyceride use during exercise (arbitrary units) | Up to 12 months
  Does exercising in the overnight-fasted state promote greater breakdown of intramuscular fat than performing exercise in the fed state?

SECONDARY OUTCOMES:
Gene expression | Up to 12 months
  The influence of pre- versus post-exercise feeding on the expression of genes related to exercise. training adaptation. Accordingly, muscle samples will be analysed using qPCr for expression of genes (relative mRNA) involved in fat metabolism (FAT/CD36, CPT1, βHAD), mitochondrial biogenesis (PGC-1α) and substrate oxidation (COXIV, CYT C, CS, SDH).

REFERENCES:
- [Derived] Edinburgh RM, Bradley HE, Abdullah NF, Robinson SL, Chrzanowski-Smith OJ, Walhin JP, Joanisse S, Manolopoulos KN, Philp A, Hengist A, Chabowski A, Brodsky FM, Koumanov F, Betts JA, Thompson D, Wallis GA, Gonzalez JT. Lipid Metabolism Links Nutrient-Exercise Timing to Insulin Sensitivity in Men Classified as Overweight or Obese. J Clin Endocrinol Metab. 2020 Mar 1;105(3):660-76. doi: 10.1210/clinem/dgz104. PMID 31628477